CLINICAL TRIAL: NCT00961922
Title: The Efficacy of Neurofeedback to Improve Processing Speed, Attention and Memory in Childhood Brain Tumour Survivors: a Randomized Controlled Trial
Brief Title: Pediatric Research on Improving Speed, Memory and Attention
Acronym: PRISMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Martha A. Grootenhuis, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UVA 2008-4013; MEC 09/137
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Brain Tumors
Keywords: childhood brain tumour survivors
MeSH Terms: conditions — Brain Neoplasms | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neurofeedback (Experimental): Children in this group receive 30 sessions of neurofeedback
  Interventions: Other: Neurofeedback
- Placebo feedback (Sham Comparator): The children in this group receive 30 sessions of placebo feedback, based on muscular tension.
  Interventions: Other: Placebo feedback
- Siblings (No Intervention): The siblings will be tested 1 time, they will function as a healthy control group.

INTERVENTIONS:
Other: Neurofeedback — 30 sessions of neurofeedback will be given twice a week at the child's home. It will take about 15 weeks to complete the training.
  Arms: Neurofeedback
Other: Placebo feedback — Feedback based on a random signal generator and muscular tension instead of brain activity. 30 sessions at home, twice a week, total 15 weeks.
  Arms: Placebo feedback

SUMMARY:
Introduction:

The aim of this study is to investigate the efficacy of neurofeedback (NFB) to improve attention, memory and processing speed in children treated for a Brain Tumour (BT). In the Netherlands every year approximately 100 children are diagnosed with a BT. Nowadays over 65% of these children have a 5-year survival. Treatment for a BT consists of neurosurgery and / or local or craniospinal radiation and / or adjuvant chemotherapy. Neurotoxicity caused by radiotherapy and / or chemotherapy (especially methotrexate) is a major cause of neurocognitive decline in Childhood Brain Tumour Survivors (CBTS).

Approach:

Studies have shown that NFB has the capacity to improve the brain systems mediating selective attention and response inhibition in children with Attention Deficit/Hyperactive Disorder (ADHD). The effectiveness is reported as comparable to methylphenidate (Ritalin) without side effects of medication. CBTS exhibit symptoms comparable to those of children with ADHD and positive response to methylphenidate has been found in CBTS. However, NFB has not been used as an intervention in CBTS yet. The effectiveness of NFB in children treated for a BT will be investigated in a randomized controlled trial. The intervention group of 30 patients will receive approximately 30 sessions of NFB; the control group will receive 30 session of placebo neurofeedback. Neuropsychological tests will be used to evaluate pre- and post-NFB intervention as well as at a 6-month follow-up.

Relevance:

If NFB proofs to be effective for CBTS this will be a great improvement for their (neuro-) psychological functioning and quality of life, without the disadvantage of the side effects of medication. The implementation of this intervention might increase cognitive and social functioning and thus facilitate integration of these children in society during childhood and school carrier as well as in adult life.

ELIGIBILITY:
Inclusion Criteria:

* Being treated for a brain tumour before the age of 16 years
* Age between 8-18 years at time of enrolment
* Off treatment at least two years
* Problems on attention, or memory or speed processing as reported by parents in screening test
* Being able to speak and understand the Dutch language

Exclusion Criteria:

* Premorbid AD/HD
* Mental or physical condition that make the neuropsychological assessment impossible to finish

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-10 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive functioning | Before (T0) and after (T1) NFB training and 6 months follow up (T2)

SECONDARY OUTCOMES:
psychosocial functioning | T0, T1 and T2

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre - UvA, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] de Ruiter MA, Schouten-Van Meeteren AY, van Mourik R, Janssen TW, Greidanus JE, Oosterlaan J, Grootenhuis MA. Neurofeedback to improve neurocognitive functioning of children treated for a brain tumor: design of a randomized controlled double-blind trial. BMC Cancer. 2012 Dec 6;12:581. doi: 10.1186/1471-2407-12-581. PMID 23217162